CLINICAL TRIAL: NCT01000649
Title: Infusion Proof-of-concept Trial Investigating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ascending Doses of FE 202158 in Patients With Vasodilatory Hypotension in Early Septic Shock
Brief Title: Effects of the V1a Agonist FE 202158 in Patients With Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FE 202158 CS02; EudraCT: 2009-010798-19
Record Dates: First submitted 2009-09-30; First posted 2009-10-23 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Septic Shock
Keywords: V1a agonist
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FE 202158 1.25 (Experimental): Patients in the arm received an intravenous infusion for up to 7 days of FE 202158 at an initial rate of 1.25 ng/kg/min.
  FE 202158 was provided as an isotonic acetate buffered stock solution of pH 4.0 in vials appropriately diluted with isotonic saline prior to use.
  Interventions: Drug: FE 202158 1.25
- FE 202158 2.5 (Experimental): Patients in the arm received an intravenous infusion for up to 7 days of FE 202158 at an initial rate of 2.5 ng/kg/min.
  FE 202158 was provided as an isotonic acetate buffered stock solution of pH 4.0 in vials appropriately diluted with isotonic saline prior to use.
  Interventions: Drug: FE 202158 2.5
- FE 202158 3.75 (Experimental): Patients in the arm received an intravenous infusion for up to 7 days of FE 202158 at an initial rate of 3.75 ng/kg/min.
  FE 202158 was provided as an isotonic acetate buffered stock solution of pH 4.0 in vials appropriately diluted with isotonic saline prior to use.
  Interventions: Drug: FE 202158 3.75
- PLCBO (Placebo Comparator): Patients in the arm received an intravenous infusion for up to 7 days of placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FE 202158 1.25 — FE 202158 at dose 1.25 ng/kg/min infused.
  Arms: FE 202158 1.25
Drug: FE 202158 2.5 — FE 202158 at dose 2.5 ng/kg/min infused.
  Arms: FE 202158 2.5
Drug: FE 202158 3.75 — FE 202158 at dose 3.75 ng/kg/min infused.
  Arms: FE 202158 3.75
Other: Placebo — Isotonic saline infused.
  Arms: PLCBO

SUMMARY:
The purpose of this trial was to examine the safety and tolerability, pharmacokinetics of FE 202158 and to assess whether it can stabilize blood pressure and reduce vascular (blood vessel) leakage. FE 202158 had previously been tested in healthy volunteers.

DETAILED DESCRIPTION:
This was a multi-centre, double-blind, randomized, placebo-controlled, parallel group trial investigating the safety, tolerability, pharmacokinetics, and pharmacodynamics of FE 202158 (using three ascending doses) in patients with vasodilatory hypotension in early septic shock, when given as continuous infusion for up to 7 days.

The trial comprised of three treatment arms where FE 202158 was administered in 1.25 ng, 2.5 ng and 3.75 ng dose, respectively. A placebo arm was also included in the trial where patients received isotonic saline.

Efficacy of FE 202158 was determined by evaluating its ability to maintain mean arterial pressure (MAP) >60 mmHg and its modulating effect on inflammatory markers. Effects of FE 202158 on other variables like vital signs, morbidity, mortality and pulmonary function were also determined.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form by the patient or a legal representative according to local regulations
* Man or woman 18 years of age or older
* Proven or suspected infection
* Low blood pressure
* Signs of decreased circulation in the tissues
* Willing to use an adequate barrier method or hormonal method of contraception, if not abstinent, from the day of informed consent to one week after the end of infusion of study medication.

Exclusion Criteria:

* Present or a history (within the last 5 years) of acute coronary syndrome (myocardial infarction or unstable angina). Patients who have been asymptomatic for 6 months after coronary revascularisation are eligible.
* Hypovolaemia suspected on clinical grounds, e.g. cold extremities with delayed capillary filling, low cardiac filling pressure, marked systolic or pulse pressure variation or positive leg raising test.
* Known or suspected cardiac failure
* Pregnancy or breastfeeding
* Any cause of hypotension other than early septic shock
* Use of vasopressin or terlipressin for blood pressure support during the current hospital admission
* Proven or suspected acute mesenteric ischemia, as judged by the investigator
* Known episode of septic shock within 1 month prior to randomisation
* Underlying chronic heart disease
* Traumatic brain injury
* Present hospitalisation with burn injury
* Symptomatic peripheral vascular disease including Raynaud's syndrome
* Previously randomized in this trial
* Intake of an investigational drug within the last 3 months (or longer if judged by the Investigator to possibly influence the outcome of the current study)
* Known participation in another clinical trial
* Considered by the investigator to be unsuitable to participate in the trial for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (16):
- United States (6):
  - Christiana Care Health System, Newark, Delaware
  - Baystate Medical Center, Springfield, Massachusetts
  - Division of Education and Research SMDC Health System, Duluth, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Baylor College of Medicine, Houston, Texas
- Belgium (4):
  - Clinique Universitaire St-Luc, Brussels
  - Erasme Hospital (Free University of Brussels), Brussels
  - University Hospital Vrije Universiteit, Brussels
  - Service des Soins Intensits, Dinant
- Canada (2):
  - Royal Columbian Hospital, Vancouver
  - St. Paul´s Hospital, Vancouver
- Denmark (4):
  - Bispebjerg Hospital, Bispebjerg
  - Rigshospitalet, Copenhagen
  - Hillerød Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre

REFERENCES:
- [Result] Russell JA, Vincent JL, Kjolbye AL, Olsson H, Blemings A, Spapen H, Carl P, Laterre PF, Grundemar L. Selepressin, a novel selective vasopressin V1A agonist, is an effective substitute for norepinephrine in a phase IIa randomized, placebo-controlled trial in septic shock patients. Crit Care. 2017 Aug 15;21(1):213. doi: 10.1186/s13054-017-1798-7. PMID 28807037
- [Derived] Rehberg S, Yamamoto Y, Sousse L, Bartha E, Jonkam C, Hasselbach AK, Traber LD, Cox RA, Westphal M, Enkhbaatar P, Traber DL. Selective V(1a) agonism attenuates vascular dysfunction and fluid accumulation in ovine severe sepsis. Am J Physiol Heart Circ Physiol. 2012 Nov 15;303(10):H1245-54. doi: 10.1152/ajpheart.00390.2012. Epub 2012 Sep 7. PMID 22961865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 55 patients were screened and 53 were randomized. One patient randomized to placebo died before dosing, and one patient randomized to 2.5 ng/kg/min was erroneously dosed with placebo.
Groups:
- FE 202158 3.75: Patients in the arm received an intravenous infusion for up to 7 days of FE 202158 at an initial rate of 3.75 ng/kg/min.The two patients randomized to FE 202158 3.75 ng group were excluded from the efficacy evaluation since meaningful analyses were not possible.
  FE 202158 was provided as an isotonic acetate buffered stock solution of pH 4.0 in vials appropriately diluted with isotonic saline prior to use.
Period: Overall Study
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | FE 202158 3.75 | PLCBO
Started | 10 (This represents Full Analysis Set population, which comprised of all dosed patients.) | 19 (This represents Full Analysis Set population, which comprised of all dosed patients.) | 2 (This represents Full Analysis Set population, which comprised of all dosed patients.) | 21 (This represents Full Analysis Set population, which comprised of all dosed patients.)
Intention-to-Treat (ITT) Analysis Set | 10 (ITT population comprised of all randomized patients.) | 20 (ITT population comprised of all randomized patients.) | 2 (ITT population comprised of all randomized patients.) | 21 (ITT population comprised of all randomized patients.)
Completed | 5 | 16 | 0 | 15
Not Completed | 5 | 3 | 2 | 6
Not completed — Adverse Event | 5 | 1 | 2 | 4
Not completed — Lost to Follow-up | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis population consist of FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | FE 202158 3.75 | PLCBO | Total
Number analyzed (Participants) | 10 | 19 | 2 | 21 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (19.6) | 57.1 (15.4) | 69 (12.7) | 63.2 (18) | 60.4 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 1 | 6 | 23
  Male | 3 | 10 | 1 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 19 | 2 | 20 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 10 | 18 | 2 | 20 | 50
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kilogram] | 64.8 (14.3) | 87.6 (28.6) | 77.5 (17.7) | 75.1 (15.3) | 77.8 (22.2)
Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: Score on a scale] — The SOFA score, is used to track a patient's status during the stay in an intensive care unit. This scoring system is used to determine the extent of a person's organ function or rate of failure. The scoring system comprise of scores for six different system: Respiratory System; Nervous System; Cardiovascular System; Liver; Coagulation; and Renal System. Score for each system ranges from 0-4 (0=normal, 4=worst)..
  Total SOFA score is a sum of the individual system score and range from 0 to 24, 0 being the better and 24 being the worst patient status.
  Score on a scale | 9.3 (2.16) | 11.2 (3.73) | 12 (0) | 10.4 (3.46) | 10.5 (3.31)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Maintaining Target Mean Arterial Pressure (MAP) (>60 mmHg) With no Open Label NE (Norepinephrine)
Description: Data were evaluated for target MAP of ≥ 60 mmHg. A 95% confidence interval (CI) was calculated and presented using Clopper-Pearson method.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of Full Analysis Set, which comprised of all patients who were dosed.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Percentage of patients
  Day 1 - 12 hrs | 0.0 [0.0 to 30.8] | 47.1 [23.0 to 72.2] | 0.0 [0.0 to 16.8]
  Day 1 - 24 hrs | 10.0 [0.3 to 44.5] | 68.8 [41.3 to 89.0] | 20.0 [5.7 to 43.7]
  Day 2 - 48 hrs | 55.6 [21.2 to 86.3] | 66.7 [38.4 to 88.2] | 38.9 [17.3 to 64.3]
  Day 4 - 96 hrs | 75.0 [34.9 to 96.8] | 66.7 [29.9 to 92.5] | 70.6 [44.0 to 89.7]
  Day 7 - 168 hrs | 62.5 [24.5 to 91.5] | 80.0 [44.4 to 97.5] | 100.0 [78.2 to 100.0]

2. Primary Outcome: Proportion of Patients Maintaining Target MAP (>60) Irrespective of Open Label NE
Description: as for outcome 1
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of Full Analysis Set, which comprised of all patients who were dosed.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Percentage of patients
  Day 1 - 12 hrs | 100.0 [63.1 to 100.0] | 100.0 [80.5 to 100.0] | 94.7 [74.0 to 99.9]
  Day 1 - 24 hrs | 87.5 [47.3 to 99.7] | 100.0 [78.2 to 100.0] | 100.0 [83.2 to 100.0]
  Day 2 - 48 hrs | 100.0 [66.4 to 100.0] | 100.0 [76.8 to 100.0] | 100.0 [81.5 to 100.0]
  Day 4 - 96 hrs | 100.0 [63.1 to 100.0] | 100.0 [63.1 to 100.0] | 100.0 [80.5 to 100.0]
  Day 7 - 168 hrs | 62.5 [24.5 to 91.5] | 100.0 [66.4 to 100.0] | 100.0 [78.2 to 100.0]

3. Primary Outcome: Cumulative Dose of Open Label NE.
Description: Cumulative Dose of Open Label NE over 7 days.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of Full Analysis Set, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: µg/kg
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
µg/kg
  Day 1 - 1 hour | 14.3 (11.6) | 13.1 (12.6) | 19.2 (14.6)
  Day 1 - 3 hours | 40.5 (35) | 30 (33.1) | 57.2 (44)
  Day 1 - 6 hours | 75.8 (60.4) | 46.9 (59.4) | 110 (84)
  Day 1 - 12 hours | 130 (96.3) | 66.5 (102) | 206 (159)
  Day 1 - 24 hours | 211 (147) | 101 (193) | 360 (270)
  Day 2 - 36 hours | 282 (206) | 122 (253) | 477 (363)
  Day 2 - 48 hours | 349 (303) | 138 (297) | 554 (445)
  Day 3 - 60 hours | 389 (377) | 150 (334) | 606 (509)
  Day 3 - 72 hours | 420 (432) | 160 (364) | 646 (567)
  Day 4 - 84 hours | 443 (471) | 169 (395) | 680 (623)
  Day 4 - 96 hours | 465 (507) | 179 (430) | 707 (674)
  Day 5 - 108 hours | 349 (342) | 186 (452) | 728 (713)
  Day 5 - 120 hours | 374 (410) | 193 (467) | 749 (757)
  Day 6 - 132 hours | 404 (474) | 200 (495) | 767 (793)
  Day 6 - 144 hours | 421 (519) | 217 (563) | 782 (823)
  Day 7 - 156 hours | 444 (582) | 236 (643) | 798 (853)
  Day 7 - 168 hours | 477 (673) | 245 (678) | 824 (897)

4. Secondary Outcome: Pharmacokinetic (PK) Parameter in Patients : Steady State Concentration
Description: PK parameters were calculated using nonlinear 2-compartment population PK model with random patient effects on clearance and volume of distribution.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FE 202158 1.25 | FE 202158 2.5
Number analyzed (Participants) | 10 | 17
ng/mL | 0.50 (0.13) | 0.99 (0.32)

5. Secondary Outcome: PK Parameter in Patients : Time to Steady State
Description: as for outcome 4
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | FE 202158 1.25 | FE 202158 2.5
Number analyzed (Participants) | 10 | 17
Hour | 7.6 (2.8) | 7.0 (2.3)

6. Secondary Outcome: PK Parameter in Patients : Clearance
Description: as for outcome 4
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Litre/hour
Arm/Group | FE 202158 1.25 | FE 202158 2.5
Number analyzed (Participants) | 10 | 17
Litre/hour | 10.0 (2.8) | 13.1 (2.9)

7. Secondary Outcome: PK Parameter in Patients : Steady State Volume of Distribution
Description: as for outcome 4
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | FE 202158 1.25 | FE 202158 2.5
Number analyzed (Participants) | 10 | 17
Litre | 25.5 (10.6) | 31.2 (14.7)

8. Secondary Outcome: PK Parameter in Patients : Initial Elimination Half-life
Description: as for outcome 4
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | FE 202158 1.25 | FE 202158 2.5
Number analyzed (Participants) | 10 | 17
Hour | 0.18 (0.09) | 0.17 (0.06)

9. Secondary Outcome: PK Parameter in Patients : Terminal Elimination Half-life
Description: as for outcome 4
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | FE 202158 1.25 | FE 202158 2.5
Number analyzed (Participants) | 10 | 17
Hour | 2.5 (1.1) | 2.7 (1.2)

10. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: The change from Baseline in CRP levels were analysed and presented as per the planned time points.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
mg/L
  Day 1 (0-24 hours) | 9.81 (42.2) | -4.84 (38.5) | 32.7 (63.8)
  Day 2 (24-48 hours) | -16.2 (89.4) | -52.4 (70.1) | -5.63 (118)
  Day 4 (72-96 hours) | -95.8 (97.1) | -176 (208) | -71.8 (97.5)
  Day 7 (144-168 hours) | -93.3 (58) | -211.0 (223) | -141 (221)

11. Secondary Outcome: Change From Baseline in Tumor Necrosis Factor (TNF)-Alpha
Description: The change from Baseline in TNF-alpha levels were analysed and presented as per the planned time points.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 1, Day 2, Day 4, and Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
ng/L
  Day 1 (0-24 hours) | -0.75 (2.37) | -0.194 (0.825) | -0.125 (0.559)
  Day 2 (24-48 hours) | -0.75 (2.37) | 0.0 (0.0) | 0.0 (0.0)
  Day 4 (72-96 hours) | -0.833 (2.5) | 0.75 (3.0) | -0.125 (0.559)
  Day 7 (144-168 hours) | -1.25 (3.06) | 1.14 (4.28) | 0.25 (0.845)

12. Secondary Outcome: Change From Baseline in Interleukin-6 (IL-6)
Description: The change from Baseline in IL-6 levels were analysed and presented as per the planned time points.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 1, Day 2, Day 4, and Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
ng/L
  Day 1 (0-24 hours) | -329 (736) | -524 (2255) | -529 (1750)
  Day 2 (24-48 hours) | -720 (1178) | -888 (1798) | -398 (2101)
  Day 4 (72-96 hours) | -794 (1206) | -1209 (1844) | -1140 (1944)
  Day 7 (144-168 hours) | -883 (1559) | -1184 (1801) | -814 (1823)

13. Secondary Outcome: Change From Baseline in Interleukin-10 (IL-10)
Description: The change from Baseline in IL-10 levels were analysed and presented as per the planned time points.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 1, Day 2, Day 4, and Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
ng/L
  Day 1 (0-24 hours) | -19.2 (54.6) | -58.3 (179) | -25.8 (51.7)
  Day 2 (24-48 hours) | -34 (70.4) | -78.9 (189) | -43 (76.1)
  Day 4 (72-96 hours) | -31.9 (95.2) | -92.3 (213) | -56.6 (84.5)
  Day 7 (144-168 hours) | 8 (24.3) | -91.7 (220) | -52.8 (97.1)

14. Primary Outcome: Infusion Rates of Open Label NE.
Description: Mean open label NE infusion rate within each predefined time period.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: µg/kg/min
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
µg/kg/min
  Day 1 - 1 hour | 0.24 (0.19) | 0.22 (0.21) | 0.32 (0.24)
  Day 1 - 3 hours | 0.22 (0.19) | 0.11 (0.17) | 0.31 (0.24)
  Day 1 - 6 hours | 0.18 (0.15) | 0.09 (0.15) | 0.28 (0.22)
  Day 1 - 12 hours | 0.13 (0.11) | 0.06 (0.14) | 0.26 (0.20)
  Day 1 - 24 hours | 0.09 (0.08) | 0.04 (0.11) | 0.19 (0.17)
  Day 2 - 36 hours | 0.10 (0.12) | 0.02 (0.07) | 0.13 (0.14)
  Day 2 - 48 hours | 0.08 (0.16) | 0.02 (0.06) | 0.08 (0.13)
  Day 3 - 60 hours | 0.03 (0.05) | 0.02 (0.06) | 0.07 (0.11)
  Day 3 - 72 hours | 0.04 (0.08) | 0.01 (0.04) | 0.05 (0.10)
  Day 4 - 84 hours | 0.03 (0.07) | 0.02 (0.06) | 0.04 (0.11)
  Day 4 - 96 hours | 0.03 (0.07) | 0.01 (0.05) | 0.03 (0.10)
  Day 5 - 108 hours | 0.0 (0.0) | 0.01 (0.01) | 0.04 (0.08)
  Day 5 - 120 hours | 0.02 (0.07) | 0.01 (0.04) | 0.03 (0.07)
  Day 6 - 132 hours | 0.02 (0.05) | 0.01 (0.04) | 0.02 (0.06)
  Day 6 - 144 hours | 0.03 (0.08) | 0.03 (0.13) | 0.02 (0.06)
  Day 7 - 156 hours | 0.04 (0.12) | 0.02 (0.08) | 0.02 (0.06)
  Day 7 - 168 hours | 0.05 (0.15) | 0.02 (0.05) | 0.01 (0.03)

15. Secondary Outcome: Change From Baseline in Interleukin-1 Receptor (IL-1R) Antagonist
Description: The change from Baseline in IL-1R levels were analysed and presented as per the planned time points.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 1, Day 2, Day 4, and Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
µg/L
  Day 1 (0-24 hours) | 0.763 (5.39) | -3.71 (7.61) | -3.28 (5.79)
  Day 2 (24-48 hours) | -3.65 (9.89) | -4.77 (10.7) | -3.84 (7.86)
  Day 4 (72-96 hours) | -6.38 (12) | -6.44 (12) | -4.51 (8.63)
  Day 7 (144-168 hours) | -3.5 (5.72) | -5.3 (10.4) | -3.9 (8.35)

16. Secondary Outcome: Change From Baseline in Heart Rate
Description: The change from Baseline in heart rate was analysed and presented as per the planned time points.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of Safety Analysis Set, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Beats per minute
  Day 1 - 3 hours | -5.7 (8.06) | -11.0 (14.1) | -4.9 (14.3)
  Day 1 - 6 hours | -4.9 (6.06) | -11.9 (14.9) | -6.55 (13.1)
  Day 1 - 9 hours | -7.2 (7.02) | -11.6 (17.3) | -5.35 (17.7)
  Day 1 - 12 hours | -7.6 (10.4) | -11.5 (13.8) | -8.45 (16.3)
  Day 1 - 15 hours | -8.6 (7.76) | -13.2 (15.5) | -4.5 (18.5)
  Day 1 - 18 hours | -7.22 (9.58) | -6.26 (19.1) | -6.95 (18.8)
  Day 1 - 21 hours | -10 (9.31) | -9.79 (14.8) | -3.2 (22.9)
  Day 1 - 24 hours | -7.44 (17.9) | -2.95 (25.1) | -2.37 (29.4)
  Day 2 - 27 hours | -7.6 (14.5) | -9.16 (19.3) | -5.4 (27.9)
  Day 2 - 30 hours | -10.3 (14.4) | -13.1 (17.4) | -7.35 (22.9)
  Day 2 - 33 hours | -9.3 (13.9) | -11.1 (15) | -10.5 (22.2)
  Day 2 - 36 hours | -6.9 (15.5) | -9.47 (16.0) | -9.05 (26.7)
  Day 2 - 39 hours | -6.7 (12.8) | -9.21 (18.4) | -7.2 (25.7)
  Day 2 - 42 hours | -6 (12.4) | -11.3 (16.5) | -9.5 (24.4)
  Day 2 - 45 hours | -1.9 (8.91) | -9.11 (14.1) | -6.5 (28.1)
  Day 2 - 48 hours | -9.9 (13.8) | -7.39 (13) | -8.9 (25)
  Day 3 - 51 hours | -10.2 (8.53) | -8.06 (16.7) | -9.11 (27.9)
  Day 3 - 54 hours | -6.11 (10.1) | -10.5 (18.1) | -9.94 (27)
  Day 3 - 57 hours | -3.67 (10.4) | -6.87 (21.8) | -7.94 (28.6)
  Day 3 - 60 hours | -1.6 (7.96) | -8.25 (22.3) | -9.4 (25.5)
  Day 3 - 63 hours | -6.78 (10.6) | -10.3 (22.6) | -10.6 (24.7)
  Day 3 - 66 hours | -5.11 (10.9) | -9.63 (19.4) | -10.9 (25)
  Day 3 - 69 hours | -9.44 (11.9) | -4.64 (24.6) | -8.35 (26.2)
  Day 3 - 72 hours | -11.9 (10.5) | -10.7 (19.8) | -8.41 (28.7)
  Day 4 - 78 hours | -2.11 (20.9) | -10.1 (18.9) | -7.06 (29.7)
  Day 4 - 84 hours | -2.4 (16.8) | -12.5 (17.6) | -9.5 (27)
  Day 4 - 90 hours | -7.38 (15.3) | -10.6 (19.2) | -4.18 (31.0)
  Day 4 - 96 hours | -2.56 (22.3) | -12.2 (16.1) | -7.78 (28)
  Day 5 - 102 hours | 4.63 (23.2) | -9.38 (19.8) | -9.65 (28.4)
  Day 5 - 108 hours | 2.11 (15.7) | -10.5 (15.9) | -6.05 (27.8)
  Day 5 - 114 hours | 1.25 (18.9) | -10.3 (16.7) | -6.12 (30.3)
  Day 5 - 120 hours | 4.11 (18.1) | -7.15 (17.4) | -5.06 (28.1)
  Day 6 - 126 hours | -0.714 (13) | -5.79 (20.2) | -4.19 (24.4)
  Day 6 - 132 hours | 1.13 (14.8) | -9.93 (16.7) | -4.22 (24.7)
  Day 6 - 138 hours | -3 (9.92) | -10.6 (14.6) | -6.4 (23.6)
  Day 6 - 144 hours | 1.38 (8.19) | -10.7 (17.3) | 1.28 (18.6)
  Day 7 - 150 hours | 0.2 (13.4) | -6 (22.3) | -1.88 (28.2)
  Day 7 - 156 hours | 6 (20.2) | -4.58 (19.9) | -8.83 (15.2)
  Day 7 - 162 hours | 6.33 (22) | -3.5 (19.1) | -11.5 (15.9)
  Day 7 - 168 hours | 8.17 (13.7) | -6.27 (21.3) | -6.94 (15.6)

17. Secondary Outcome: Change From Baseline in Fluid Balance
Description: The change from Baseline in fluid balance were analysed and presented as per the planned time points. The fluid balance was adjusted for length of time interval and weight.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: mL/hour/kg
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
mL/hour/kg
  Day 1 - 0-6 hours | -2.11 (6.99) | -0.0513 (3.08) | -0.477 (2.03)
  Day 1 - 0-12 hours | -3.56 (6.34) | -0.889 (3.29) | -0.578 (2.2)
  Day 1 - 12-18 hours | -3.66 (6.68) | -1.41 (3.11) | -0.98 (2.42)
  Day 1 - 18-24 hours | -3.49 (6.78) | -1.47 (3.45) | -0.119 (2.95)
  Day 2 - 24-30 hours | -3.49 (5.56) | -1.75 (3.1) | -0.905 (2.68)
  Day 2 - 30-36 hours | -3.42 (5.63) | -0.963 (3.82) | -1.47 (3.04)
  Day 2 - 36-42 hours | -3.34 (6.09) | -1.82 (3.36) | -2.54 (3.48)
  Day 2 - 42-48 hours | -3.82 (6.66) | -2.18 (3.51) | -2.01 (3.52)
  Day 3 - 48-54 hours | -3.2 (6.26) | -1.97 (3.68) | -1.93 (2.59)
  Day 3 - 54-60 hours | -4.42 (7.6) | -2.85 (3.52) | -2.91 (2.55)
  Day 3 - 60-66 hours | -4.31 (6.68) | -2.86 (3.33) | -2.21 (2.54)
  Day 3 - 66-72 hours | -4.64 (6.71) | -2.75 (3.76) | -2.54 (2.79)
  Day 4 - 72-84 hours | -4.82 (6.47) | -2.52 (3.36) | -2.35 (3.28)
  Day 4 - 84-96 hours | -4.01 (6.08) | -2.4 (3.55) | -2.67 (3.58)
  Day 5 - 96-108 hours | -4.3 (6.08) | -2.84 (4.08) | -2.62 (3.2)
  Day 5 - 108-120 hours | -4.12 (5.99) | -3.3 (3.84) | -2.22 (2.78)
  Day 6 - 120-132 hours | -4.17 (6.19) | -3.04 (3.86) | -2.67 (3.45)
  Day 6 - 132-144 hours | -5.41 (6.62) | -2.99 (3.17) | -2.87 (3.19)
  Day 7 - 144-156 hours | -5.56 (6.34) | -2.37 (3.1) | -2.8 (2.69)
  Day 7 - 156-168 hours | -5.38 (6.09) | -2.85 (3.13) | -2.6 (2.46)

18. Secondary Outcome: SOFA Score
Description: The SOFA score, is used to track a patient's status during the stay in an intensive care unit. This scoring system is used to determine the extent of a person's organ function or rate of failure. The scoring system comprise of scores for six different system: Respiratory System; Nervous System; Cardiovascular System; Liver; Coagulation; and Renal System. Score for each system ranges from 0-4 (0=normal, 4=worst).
  Total SOFA score is a sum of the individual system score and range from 0 to 24, 0 being the better and 24 being the worst patient status.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7, Day 14 and Day 29
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Score on a scale
  Day 1 (0-24 hours) | 8.7 (2.45) | 11.9 (3.43) | 10.5 (3.22)
  Day 2 (24-48 hours) | 8.0 (3.5) | 8.68 (3.07) | 9.0 (2.83)
  Day 3 (48-72 hours) | 7.6 (3.53) | 8.32 (3.64) | 8.2 (2.57)
  Day 4 (72-96 hours) | 6.8 (3.91) | 7.5 (3.91) | 8.05 (2.82)
  Day 5 (96-120 hours) | 6.6 (4.2) | 7.06 (3.49) | 7.44 (2.77)
  Day 6 (120-144 hours) | 5.22 (3.35) | 6.63 (3.32) | 7.06 (3.02)
  Day 7 (144-168 hours) | 4.63 (3.7) | 5.93 (3.65) | 7.18 (2.65)
  Day 14 | 5.0 (4.36) | 4.27 (3.82) | 3.53 (1.81)
  Day 28 | 1.75 (2.36) | 2.7 (2.63) | 2.11 (0.93)

19. Secondary Outcome: Pulmonary Function : Change From Baseline in PaO2/FiO2
Description: Change from Baseline in PaO2/FiO2 was observed at each time-point.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of Safety Analysis Set, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Ratio
  Day 1 - 6 hours | -1.7 (80.3) | 1.35 (85.2) | -7.06 (99.9)
  Day 1 - 12 hours | 22.8 (95.3) | -11.9 (61.9) | 7.32 (72.3)
  Day 1 - 18 hours | 12.1 (86.7) | -17.6 (94) | 9.21 (88.5)
  Day 1 - 24 hours | -4.22 (84.4) | 34.8 (144) | -3.68 (92.8)
  Day 2 - 30 hours | 54.3 (142) | -16.5 (116) | 12.4 (96.1)
  Day 2 - 36 hours | 15.8 (112) | 6.89 (115) | 39.8 (100)
  Day 2 - 42 hours | 28.6 (137) | -1.27 (118) | 14.6 (123)
  Day 2 - 48 hours | 16.2 (74.3) | 10.3 (105) | 8.24 (135)
  Day 3 - 54 hours | 24.8 (137) | 49.5 (81.1) | 19.4 (129)
  Day 3 - 60 hours | 118 (172) | 9.8 (106) | 50 (108)
  Day 3 - 66 hours | 64.7 (131) | 6.38 (70.1) | 17.7 (120)
  Day 3 - 72 hours | 51.7 (120) | 74.2 (89.8) | 21.8 (119)
  Day 4 - 84 hours | 61.4 (115) | 7.54 (85.4) | 44.1 (97.9)
  Day 4 - 96 hours | 96.1 (97.2) | 65.5 (112) | 22.9 (128)
  Day 5 - 108 hours | 123 (233) | 30.1 (49.3) | 38.4 (115)
  Day 5 - 120 hours | 63.7 (130) | 5.89 (58.3) | 51.8 (132)
  Day 6 - 132 hours | 123 (154) | 7.17 (89.6) | 40.3 (133)
  Day 6 - 144 hours | 42.8 (69.3) | 30.2 (83.7) | -19.6 (114)
  Day 7 - 156 hours | 37.6 (68.3) | 40.9 (83.8) | -19.1 (151)
  Day 7 - 168 hours | 117 (255) | 59 (68.1) | -30.2 (105)

20. Secondary Outcome: Pulmonary Function : Change From Baseline in Tidal Volume
Description: Change from Baseline in tidal volume was observed at each time-point.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of Safety Analysis Set, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
mL/kg
  Day 1 - 6 hours | -0.533 (0.666) | 0.196 (0.736) | -0.0189 (1.91)
  Day 1 - 12 hours | -0.208 (0.708) | 0.256 (0.794) | -0.24 (1.37)
  Day 1 - 18 hours | 0.171 (0.957) | 0.141 (0.539) | -0.26 (1.17)
  Day 1 - 24 hours | -1.1 (1.16) | 0.285 (1.02) | 0 (1.64)
  Day 2 - 30 hours | -0.81 (1.15) | 0.34 (1.46) | -0.0259 (2.11)
  Day 2 - 36 hours | -0.208 (1.24) | 0.145 (0.734) | -0.223 (1.64)
  Day 2 - 42 hours | -0.478 (1.13) | 0.298 (1.21) | -1.19 (1.33)
  Day 2 - 48 hours | -0.604 (1.52) | 0.532 (1.31) | -0.538 (2.02)
  Day 3 - 54 hours | -0.118 (1.86) | 0.163 (1.19) | -0.859 (1.84)
  Day 3 - 60 hours | -0.214 (1.1) | 0.62 (1.69) | -0.951 (1.57)
  Day 3 - 66 hours | -0.01 (1.37) | 0.628 (1.25) | -0.592 (1.98)
  Day 3 - 72 hours | -0.23 (1.49) | 1.48 (3.19) | -0.348 (1.78)
  Day 4 - 84 hours | 0.966 (2.44) | 0.466 (1.89) | -0.844 (2.03)
  Day 4 - 96 hours | -0.528 (1.62) | -0.313 (0.864) | -1.16 (2.44)
  Day 5 - 108 hours | 0.633 (1.93) | 0.207 (1.39) | -0.723 (2.14)
  Day 5 - 120 hours | -0.338 (2.24) | -0.412 (0.709) | -0.613 (1.73)
  Day 6 - 132 hours | -0.298 (1.41) | 0.462 (1.86) | -0.746 (1.41)
  Day 6 - 144 hours | -0.458 (1.09) | 0.292 (2.69) | -0.823 (1.71)
  Day 7 - 156 hours | 0.483 (1.13) | -0.733 (1.32) | -2.14 (2.53)
  Day 7 - 168 hours | -0.0667 (1.1) | -0.438 (1.37) | -2.19 (2.93)

21. Secondary Outcome: Change From Baseline in Arterial Blood Gas (Lactate)
Description: Change from Baseline in arterial blood gas (lactate) was observed at each time-point.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of Safety Analysis Set, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
mmol/L
  Day 1 - 6 hours | 0 (0.482) | -0.367 (1.03) | -0.0278 (0.647)
  Day 1 - 12 hours | -0.489 (0.857) | -0.833 (1.53) | -0.0444 (0.912)
  Day 1 - 18 hours | -0.525 (0.932) | -1.01 (1.66) | -0.3 (0.974)
  Day 1 - 24 hours | -0.9 (1.06) | -1.01 (1.93) | -0.533 (1.13)
  Day 2 - 30 hours | -0.975 (1.09) | -1.33 (2.5) | -0.647 (1.12)
  Day 2 - 36 hours | -0.744 (1.01) | -1.45 (2.57) | -0.683 (1.19)
  Day 2 - 42 hours | -0.844 (0.958) | -1.57 (2.84) | -0.917 (1.11)
  Day 2 - 48 hours | -0.722 (1.11) | -1.68 (2.84) | -0.888 (1.29)
  Day 3 - 54 hours | -0.788 (1.22) | -1.6 (1.99) | -1.11 (1.33)
  Day 3 - 60 hours | -0.163 (1.13) | -1.15 (1.65) | -0.925 (1.4)
  Day 3 - 66 hours | -0.371 (1.08) | -1.01 (1.84) | -1.15 (1.39)
  Day 3 - 72 hours | -0.643 (1.03) | -1.27 (1.92) | -0.879 (1.45)
  Day 4 - 84 hours | -0.5 (1.07) | -0.975 (1.76) | -1.12 (1.36)
  Day 4 - 96 hours | -0.671 (0.948) | -0.52 (0.902) | -1.34 (1.47)
  Day 5 - 108 hours | -0.633 (0.963) | -1.37 (2.07) | -1.21 (1.51)
  Day 5 - 120 hours | -0.6 (1) | -1.06 (1.89) | -1.38 (1.5)
  Day 6 - 132 hours | -0.717 (0.768) | -1.26 (1.87) | -1.23 (1.27)
  Day 6 - 144 hours | -1.03 (1.01) | -1.28 (1.84) | -1.12 (0.946)
  Day 7 - 156 hours | -0.56 (0.783) | -2.17 (3.44) | -1.3 (1.36)
  Day 7 - 168 hours | -0.533 (2.2) | -1.6 (1.92) | -1.34 (1.62)

22. Secondary Outcome: Days Alive and Free of Any Organ Dysfunction at Day 7
Description: Percentage of days alive and free of any organ dysfunction (i.e. no. of days divided by 7).
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Percentage of days | 5.38 (10.7) | 3.8 (11.4) | 0.0 (0.0)

23. Secondary Outcome: Percentage of Patients Alive and Free of All Vasopressors
Description: Percentage of patients alive and free of all vasopressors was assessed on Days 7, 14, and 28.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 7, Day 14 and Day 28
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Number; unit: Percentage of patients
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Percentage of patients
  Day 7 | 60.0 | 57.9 | 73.7
  Day 14 | 40.0 | 89.5 | 94.7
  Day 28 | 50.0 | 82.4 | 83.3

24. Secondary Outcome: Percentage of Days Alive and Free of Dialysis
Description: Percentage of days alive and free of dialysis was assessed on Days 7, 14, and 28.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 7, Day 14 and Day 28
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Percentage of days
  Day 7 | 53.9 (43.4) | 79.7 (36.4) | 83.2 (24.1)
  Day 14 | 55.1 (45.0) | 80.1 (33.4) | 87.6 (16.9)
  Day 28 | 50.5 (43.9) | 78.5 (35.4) | 88.6 (19.8)

25. Secondary Outcome: Percentage of Days Alive and Free of Ventilation
Description: Percentage of days alive and free of ventilation was assessed on Days 7, 14, and 28.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 7
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Percentage of days | 31.3 (37.5) | 53.8 (38.9) | 23.1 (34.8)

26. Secondary Outcome: Mortality
Description: Mortality was assessed as percentage of patients dead at pre-specified time points.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: At Day 1, 7, 14, and 28
Population: The analysis population consist of FAS, which comprised of all patients who were dosed.
Measure: Number; unit: Percentage of patients
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Percentage of patients
  At Day 1 | 0.0 | 0.0 | 0.0
  At Day 7 | 20.0 | 0.0 | 0.0
  At Day 14 | 40.0 | 0.0 | 0.0
  At Day 28 | 50.0 | 5.3 | 21.1

27. Secondary Outcome: Incidence of Abnormal Changes in ECG
Description: The number of patients having abnormal changes in ECG variables during the trial period was presented.
  The patients (n=2) in the FE 202158 3.75 ng/kg/min dose group were both discontinued within 5 hours after start of infusion. Therefore, no adequate data was available to perform the analysis for the outcome.
Time Frame: Day 1 up to Day 7
Population: The analysis population consist of Safety Analysis Set, which comprised of all patients who were dosed.
Measure: Number; unit: Number of patients
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | PLCBO
Number analyzed (Participants) | 10 | 19 | 21
Number of patients
  Heart rate <=50 beats per minute | 0 | 1 | 4
  Heart rate >=100 beats per minute | 5 | 11 | 8
  PQ interval <=120 msec | 1 | 6 | 5
  PQ interval >=220 msec | 0 | 0 | 1
  QRS interval >=120 msec | 2 | 2 | 4
  QT interval >=450 msec | 3 | 4 | 8
  QT interval >=480 msec | 1 | 2 | 6
  QT interval >=500 msec | 0 | 2 | 3
  QT interval >=30 msec increase from Baseline | 7 | 15 | 14
  QT interval >=60 msec increase from Baseline | 5 | 13 | 12
  QTcF >=450 msec | 1 | 9 | 10
  QTcF >=480 msec | 0 | 3 | 7
  QTcF >=500 msec | 0 | 2 | 6
  QTcF >=30 msec increase from Baseline | 3 | 14 | 11
  QTcF >=60 msec increase from Baseline | 2 | 9 | 9

ADVERSE EVENTS:
Time Frame: 28 days
Description: AE information was collected throughout the trial from the time of obtaining informed consent until the end of follow-up.
Groups:
- FE 202158 1.25: Patients in the arm received a continuous intravenous infusion of FE 202158 1.25 ng/kg/min up to seven consecutive days.
  FE 202158 was provided as an isotonic acetate buffered stock solution of pH 4.0 in vials appropriately diluted with isotonic saline prior to use.
- FE 202158 2.5: Patients in the arm received a continuous intravenous infusion of FE 202158 2.5 ng/kg/min up to seven consecutive days.
  FE 202158 was provided as an isotonic acetate buffered stock solution of pH 4.0 in vials appropriately diluted with isotonic saline prior to use.
- FE 202158 3.75: Patients in the arm received a continuous intravenous infusion of FE 202158 3.75 ng/kg/min up to seven consecutive days.
  FE 202158 was provided as an isotonic acetate buffered stock solution of pH 4.0 in vials appropriately diluted with isotonic saline prior to use.
- PLCBO: Patients in the arm received a continuous intravenous infusion of isotonic saline up to seven consecutive days.
Arm/Group | FE 202158 1.25 | FE 202158 2.5 | FE 202158 3.75 | PLCBO
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/19 | 2/2 | 6/21
Other Adverse Events (participants affected / at risk) | 6/10 | 14/19 | 0/2 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 202158 1.25 (N=10) | FE 202158 2.5 (N=19) | FE 202158 3.75 (N=2) | PLCBO (N=21)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 202158 1.25 (N=10) | FE 202158 2.5 (N=19) | FE 202158 3.75 (N=2) | PLCBO (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 7 (7)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac valve vegetation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia herpes viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood phosphorus (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida serology positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal cavity drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.